CLINICAL TRIAL: NCT03513120
Title: Return to Sport After Posterior Spinal Fusion in Adolescent Athletes With Idiopathic Scoliosis: a Prospective Study
Brief Title: Return to Sport After Posterior Spinal Fusion
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2473
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Adolescent Idiopathic Scoliosis; Posterior Spinal Fusion
Keywords: Adolescent Idiopathic Scoliosis; Posterior Spinal Fusion; Return to Sport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this prospective study is to determine when adolescent athletes with idiopathic scoliosis are able to return to sports participation after posterior spinal fusion surgery.

DETAILED DESCRIPTION:
The investigators aim to determine at what time subjects return to athletic activity, and how long after surgery they are performing at pre-surgical levels. The investigators will enroll adolescent athletes that meet the inclusion criteria below, and follow their postoperative activity level with standardized activity questionnaires on a monthly basis until the subject reaches their baseline pre-surgical performance level. The investigators primary aim is to determine at what time patients return to sports without any restrictions to contact level or type of play. The investigators secondary aim is to quantitatively assess when patients are able to compete at their prior level of play as determined by self-assessment surveys, as well as identify any post-operative complications in these patients after return to sports.

ELIGIBILITY:
Inclusion Criteria:

* Level of play: high school or club level
* Frequency of play at above level: >3mos/year
* Age: 10-18 years of age (inclusive)
* Sports: at least one sport, contact, non-contact, or collision. No sports exclusion criteria
* Spinal deformity criteria: Adolescent idiopathic scoliosis, curve size 40-75 degrees

Exclusion Criteria:

* Play at recreational/intramural level
* Non-English Speaking Patient
* Sports participation <3 mos/year
* Non idiopathic etiology or curves >75 degrees
* Treatment outside of Children's Hospital Colorado provider care network

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All enrolled subjects will be competitive athletes with a diagnosis of adolescent idiopathic scoliosis and plans to undergo posterior spinal fusion.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Return to Sport | Less than 1 year following surgery
  Identify at what time patients return to sports without any restrictions.

SECONDARY OUTCOMES:
Physical Function Levels | Less than 1 year following surgery
  Identify at what time patients report physical function returns to their pre-surgical levels.
Postoperative Complications | Up to 1 year follow up
  Identify any postoperative complications related to release to full activity one month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Garg, MD, Study Director — Children's Hospital Colorado; Allison Tetreault, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers